CLINICAL TRIAL: NCT02942459
Title: Music Therapy for Treatment of Patients Suffering From Schizophrenia With Negative Symptoms - A Double-blinded Study
Brief Title: Music Therapy Towards Schizophrenia, Negative Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inge Nygaard Pedersen (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor-Investigator, Inge Nygaard Pedersen, Ass. Professor. PhD, Aalborg Psychiatric Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N-20150054
Record Dates: First submitted 2016-09-20; First posted 2016-10-24 (Estimated); Last update posted 2019-07-08 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia
Keywords: music therapy; double-blinded; Randomized Controlled study (RCT); Schizophrenia, negative symptoms
MeSH Terms: conditions — Schizophrenia | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Music Therapy (Experimental): 25 Weekly Hours of Music Therapy adapted to the Needs of the Participants. Interventions can be Active (playing Music, singing, improvising, Song-writing) or Receptive (Listening to selected Play-lists, or to the Participants´ favored Music).
  A Manual is created and trained with the Music Therapists, which distinguishes between
  1. Unique and Essential Principles for Music Therapy with people suffering from Schizophrenia with negative Symptoms,
  2. Essential but not Unique Principles,
  3. Acceptable but not necessary Principles,
  4. Not acceptable and Proscribed Principles. These Principles concern Attitude and Listening Perspectives by the Music Therapist, how to conduct the Musical Interventions and Questions of Frames for the Music Therapy Work.
  Interventions: Other: Music therapy
- Music Listening (Active Comparator): 25 Weekly Hours of Being together with an unknown Care Staff Member listening to Music from selected Play-Lists. Music Therapists at the Music Therapy Research Clinic at Aalborg University Hospital, Psychiatry have developed Play-Lists in a Taxonomy from very Supportive to less Supportive Music including around 100 Hours of Music all together on the Lists.
  A Manual is created and trained with the Care Staff Members. Here the Activities are much more limited (only Music Listening to the Play-Lists are allowed). No Therapeutical Conversation is allowed.
  Interventions: Other: Music Listening

INTERVENTIONS:
Other: Music therapy — 25 Weekly Hours of Music Therapy by an Educated Music Therapist
  Arms: Music Therapy
Other: Music Listening — 25 weekly Hours of Being Together with an unknown Care Staff Member
  Arms: Music Listening

SUMMARY:
The Aim of this National study is to examine whether music therapy can reduce negative symptoms and raise Quality of Life for patients suffering from Schizophrenia. It is an Randomized Controlled Trial (RCT), double-blinded study with two arms. 120 Participants are anticipated. The two Arms consist of 25 weekly hours of Music Therapy by educated Music Therapists and time compensated Music Listening by unknown Care Staff Members.

The Study is a close Cooperation between Aalborg University (The Music Therapy Research Clinic) and Aalborg University Hospital, Psychiatry.

DETAILED DESCRIPTION:
Schizophrenia includes 1 % of the Population in Denmark (DK) and often ends up to be chronically. Negative Symptoms are difficult to reduce by Medication and Psychosocial Treatment Possibilities are searched for. Three Cochrane Reviews (2005, 2011, 2017) have been conducted concerning Music Therapy and Schizophrenia with Positive Results. This RCT, double-blinded Study aims at verifying, if these Results can be Recognized in the Danish Health System. It also aims at being similar to Biomedical Study Designs as much as possible to strengthen the Evidence of the Study. A Power Calculation showed, that a minimum of 44,5 Participants in each Arm should be available, but as drop out can be anticipated with this Population, 60 Participants in each Arm were recommended. The screening Procedure is Comprehensive as it aims at securing, that the negative Symptoms are part of the Illness Schizophrenia and not side Effects from Medication or simultaneous Depression (See the Inclusion- and Exclusion criteria).

The Measurement Tools are as follows:

At Baseline, after 15 Sessions and at Termination:

* The Positive and Negative Syndrome Scale (PANSS),
* Brief Negative Symptom Scale (BNSS),
* Quality of Life (WHOQOL-Bref),
* Calgary Depression Scale for Schizophrenia (CDSS),
* Board of Clinical Examinations (Danish Questionnaire) (UKU)
* Global Assessment of Functioning Scale (GAF) 4 Weeks after Termination Follow Up Interview. In the Arm of Music Therapy Audio Recording of Music Interventions are done in Session 1,15 and 25.
* Helping Alliance Questionnaire, patient version, (Haq-II) This Haq-II is filled out after 5 sessions and after 15 Sessions and at Termination together with a Research Assistant in both Arms.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years
* A Diagnosis of Schizophrenia International Classification of Diseases (ICD-10 (F20))
* The Positive and Negative Syndrome Scale (PANNS), negative subscale has to show ≥ 4 on two of the following parameters:

(N1) subdued affect, (N2) emotional withdrawal, (N3) poor contact and (N4) passive/apathetic social withdrawal.

Exclusion Criteria:

* Debut of schizophrenia less than 2 years ago.
* Patients in acute worsening of schizophrenia defined as hospitalization within the last three months.
* PANNS positive subscale (P1-P7) >28.
* Patients who have their psychotropics changed within the last months.
* Significant drug dependency conflicting participation in the study.
* Presence of secondary symptoms defined as Depression - CDSS score > 7
* Neurological side effects - UKU score > 1 in one of the following items: 2.1, 2.2, 2.3, 2.5, 2.6
* Sedative side effects - UKU item 1.3 score > 1.
* No individual music therapy within the last two months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-09-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline at 25 Sessions of Music Therapy in Negative Symptoms. Psychological Questionnaires | Up til 30 weeks
  The Positive and Negative Syndrome Scale (PANSS). Negative Subscale.

SECONDARY OUTCOMES:
Change in Quality of Life from Baseline at 25 sessions. Psychological Questionnaire | Up till 30 weeks
  Quality of Life (WHOQOL-Bref)
Functional Changes from Baseline to Termination. Psychological Questionnaire | Up to 30 weeks
  Global Assessment of Functioning (GAF)
Changes of Anhedonic Features from Baseline at 25 Sessions of Music Therapy. Psychological Questionnaire | Up to 30 weeks
  Brief negative Symptom Scale (BNSS). Anhedonic Subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Inge N. Pedersen, Ass. Prof., Principal Investigator — Aalborg University
Locations (1):
- Aalborg University Hospital, Aalborg, North Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hannibal N, Pedersen IN, Bertelsen LR, Nielsen RE, Gold C. Process-outcome relations in music therapy versus music listening for people with schizophrenia viewed through a mediational model: the role of the therapeutic alliance. Front Psychiatry. 2023 May 2;14:1120003. doi: 10.3389/fpsyt.2023.1120003. eCollection 2023. PMID 37200903
- [Derived] Pedersen IN, Bonde LO, Hannibal NJ, Nielsen J, Aagaard J, Gold C, Rye Bertelsen L, Jensen SB, Nielsen RE. Music Therapy vs. Music Listening for Negative Symptoms in Schizophrenia: Randomized, Controlled, Assessor- and Patient-Blinded Trial. Front Psychiatry. 2021 Dec 21;12:738810. doi: 10.3389/fpsyt.2021.738810. eCollection 2021. PMID 34992553